CLINICAL TRIAL: NCT02886845
Title: Study of Two Single Nucleotide Polymorphisms in Chinese Breast Cancers
Brief Title: Genotyping 2 SNPs in Chinese Breast Cancers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Song Hongping (Other)
Responsible Party: Sponsor-Investigator, Song Hongping, PhD, The First Affiliated Hospital of the Fourth Military Medical University
Organization: The First Affiliated Hospital of the Fourth Military Medical University (Other)
Other Study IDs: BRCA-Genetics-2016
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: rs185670819 and rs183489969
Keywords: SNP,Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chinese Breast Cancers: Woman with breast cancer that have been diagnosed in clinic
  Interventions: Genetic: rs183489969,rs185670819
- healthy controls: Woman without breast cancer
  Interventions: Genetic: rs183489969,rs185670819

INTERVENTIONS:
Genetic: rs183489969,rs185670819 — compare the frequency of two germline mutations in breast cancers and controls

SUMMARY:
The purpose of this study is to determine the frequency of two Single Nucleotide Polymorphisms (SNPs) by sanger-sequencing in Breast Cancers and healthy controls .

DETAILED DESCRIPTION:
Since the 1990s breast cancers incidence of china has increased more than twice as fast as global rates. Chinese patients are responsible for 12.2% of all newly diagnosed breast cancers and 9.6% of all deaths to world breast cancers. Breast cancer is now the second frequently diagnosed cancer and is the leading cause of cancer-related death in Chinese women.

Two of the most prevalent breast cancer susceptibility genes are BRCA1and BRCA2. However，because of population based Genetic heterogeneity, the frequency of BRCA1/BRCA2 mutation is not as high in Caucasian population as in China. Anyway, the mean age at diagnosis of breast cancer in China is almost 10 years younger and more cases are diagnosed before 40 than those in Caucasians. Therefore, it is believed that there are certain specific susceptibility loci in Chinese breast cancers.

In preliminary experiments, investigators found two germline mutations may associate with Chinese breast cancers.

The purpose of the study is to determine the frequency of two germline mutations by sanger-sequencing in a larger sample of Chinese breast cancers

ELIGIBILITY:
Inclusion Criteria:

* Woman aged superior to 18 years old Inform consent signed Woman without breast cancer and family history of cancer

Exclusion Criteria:

* No inform consent signed Patient under guardianship, curatorship Psychosocial disorder

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Woman aged superior to 18 years old
  * Inform consent signed
  * Woman with breast cancer that have been diagnosed in clinic
  Exclusion Criteria
  * No inform consent signed
  * Patient under guardianship, curatorship
  * Psychosocial disorder
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-08; Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Genotyping of 2 SNPs ( rs185670819 and rs183489969) in Chinese breast cancer patients and age-matched healthy control women . | January of 2019

SECONDARY OUTCOMES:
Both of the 2 SNPs' minor allele frequency or affected ratio shows statistically significant differences between case and control groups | June of 2019

CONTACTS AND LOCATIONS:
Overall Officials: hongping song, PhD, Principal Investigator — The First Affiliated Hospital of Fourth Military Medical University
Locations (1):
- The First Affiliated Hospital of Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No